CLINICAL TRIAL: NCT01625117
Title: Mental Health and Aggression in Congolese Ex-combatants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Susanne Schaal, Susanne Schaal, University of Konstanz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DFG_2011
Record Dates: First submitted 2012-01-16; First posted 2012-06-21 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Appetitive Aggression; Posttraumatic Stress Disorder
Keywords: Treatment of ex-combatants; Narrative Exposure Therapy for ex-combatants; Appetitive Aggression; Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention)
- A variant of Narrative exposure therapy (Experimental)
  Interventions: Behavioral: A variant of Narrative Exposure Therapy

INTERVENTIONS:
Behavioral: A variant of Narrative Exposure Therapy — During the proposed therapy, the client constructs a chronological narrative of his or her whole life which includes all traumatic experiences and perpetrated violent acts. All emotions, cognitions, sensory information, and physiological reactions are activated and linked to the autobiographical context.In five sessions the therapist and the client try to go through all important traumatic experiences and perpetrated violent acts. The sixth session is a group session with four to five clients. The group session is oriented on Interpersonal Psychotherapy and focuses on the role change from soldier to civilian.
  Arms: A variant of Narrative exposure therapy

SUMMARY:
The purpose of this study is examine, whether a treatment approach, which is specifically tailored for perpetrators who have participated in violence (a variant of Narrative Exposure Therapy) is effective in the reduction of instrumental aggression and symptoms of posttraumatic stress disorder.

DETAILED DESCRIPTION:
The reintegration of former child soldiers and ex-combatants is a big challenge in war-torn countries. Former child soldiers and ex-combatants often suffer from mental health problems and show enhanced levels of aggression. The present study focuses on the reduction of appetitive aggression and the improvement of mental health in former child soldiers and ex-combatants in DR Congo.

ELIGIBILITY:
Inclusion Criteria:

* Ex-combatants in Congo who live in a re-integration camp

Ages: 16 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Appetitive aggression (Appetitive Aggression Scale) | 6 months
Symptoms of posttraumatic stress disorder (Posttraumatic Diagnostic Scale, PDS) | 6 months

SECONDARY OUTCOMES:
Symptoms of depression (Mini-International Neuropsychiatric Interview) | 6 months
Functionality (Work and Social Adjustment Scale) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Elbert, Prof. Dr., Study Director — University of Konstanz
Locations (1):
- Reintegration camp for ex-combatants, Goma, Republic of the Congo